CLINICAL TRIAL: NCT04313023
Title: A Phase 2 Multiple Dose Study to Evaluate the Efficacy and Safety of PUL-042 Inhalation Solution in Reducing the Infection Rate and Progression to COVID-19 in Adults Exposed to SARS-CoV-2
Brief Title: The Use PUL-042 to Reduce the Infection Rate and Progression to COVID-19 in Adults Exposed to SARS-CoV-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmotect, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PUL-042-501
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PUL-042 Inhalation Solution (Experimental): PUL-042 Inhalation Solution given by nebulization on Study Days 1, 3, 6, and 10
  Interventions: Drug: PUL-042 Inhalation Solution
- Sterile saline for inhalation (Placebo Comparator): Sterile saline for inhalation given by nebulization on Study Days 1, 3, 6, and 10
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PUL-042 Inhalation Solution — 20.3 µg Pam2 : 29.8 µg ODN/mL (50 µg PUL-042) PUL-042 Inhalation Solution
  Arms: PUL-042 Inhalation Solution
Drug: Placebo — Sterile saline for inhalation
  Arms: Sterile saline for inhalation

SUMMARY:
Subjects who have documented exposure to SARS-CoV-2 (COVID-19) will receive 4 doses of PUL-042 Inhalation Solution or 4 doses of a placebo solution by inhalation over 10 days. Subjects will be followed for the incidence and severity of COVID-19 over 28 days. Subjects will be tested for infection with SARS-CoV-2 at the beginning, middle and end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have recent exposure to SARS-CoV-2 (such as repeated or extensive exposure to an infected individual(s) or cohabiting with a SARS-CoV-2 positive individual).
2. Subjects must be 50 years or older if the exposure is due to cohabitation.
3. Subjects must be free of clinical signs or symptoms of a potential COVID-19 diagnosis (Ordinal Scale of Clinical Improvement score of 0) with a SARS-CoV-2 infection symptom score (fever, cough, shortness of breath, and fatigue) of 0 in each category.
4. Spirometry (forced expiratory volume in one second FEV1 and forced vital capacity [FVC]) ≥70% of predicted value.
5. If female, the subject must be surgically sterile or ≥ 1 year postmenopausal. If of child-bearing potential (including being < 1years postmenopausal) and, if participating in sexual activity that may lead to pregnancy, the subject agrees to use an effective dual method of birth control (acceptable methods include intrauterine device, spermicide, barrier, male partner surgical sterilization, and hormonal contraception) during the study and through 30 days after completion of the study.
6. If female, must not be pregnant, plan to become pregnant, or nurse a child during the study and through 30 days after completion of the study. A pregnancy test must be negative at the Screening Visit, prior to dosing on Day 1.
7. If male, must be surgically sterile or, if not surgically sterile and if participating in sexual activities that may lead to pregnancy, be willing to practice two effective methods of birth control (acceptable methods include barrier, spermicide, or female partner surgical sterilization) during the study and through 30 days after completion of the study.
8. Ability to understand and give informed consent.

Exclusion Criteria:

1. Previous infection with SARS-CoV-2.
2. Receipt of any vaccine for the prevention of COVID-19 (single or multiple doses).
3. A SARS-CoV-2 infection symptom score greater than 0 in any of the 4 catergories (fever, cough, shortness of breath or fatigue) at the time of screening (Ordinal Scale for Clinical Improvement score of 0).
4. Known history of chronic pulmonary disease (e.g., asthma [including atopic asthma, exercise-induced asthma, or asthma triggered by respiratory infection], chronic pulmonary disease, pulmonary fibrosis, COPD), pulmonary hypertension, or heart failure.
5. Any condition which, in the opinion of the Principal Investigator, would prevent full participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Broom, MD, Study Director — Pulmotect, Inc.
Locations (15):
- United States (15):
  - University of California Irvine, Orange, California
  - Premier Urgent Care of California, San Bernardino, California
  - Clinical Research of South Florida Alliance for Multispecialty Research, Coral Gables, Florida
  - Invesclinic US LLC, Fort Lauderdale, Florida
  - Luminous Cinical Research- South Florida Urgent Care, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - DBC Research, Tamarac, Florida
  - Affinity Clinical Research, LLC, Tampa, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Willis-Knighton Physcian Network, Bossier City, Louisiana
  - Ascension St John, Bartlesville, Oklahoma
  - Ascension St. John, Tulsa, Oklahoma
  - Invesclinic US LLC, Edinburg, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Next Level Urgent Care, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Started | 108 | 109
Completed | 100 | 107
Not Completed | 8 | 2

BASELINE CHARACTERISTICS:
Population: A total of 217 participants were randomized to the study: 7 participants were randomized but not treated, 210 (96.8%) participants were included in the ITT (Intent-to-Treat) Population and Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation | Total
Number analyzed (Participants) | 102 | 108 | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 99 | 190
  >=65 years | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (13.64) | 45.6 (14.4) | 47.1 (14.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 120
  Male | 42 | 48 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 68 | 78 | 146
  Not Hispanic or Latino | 34 | 30 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 16 | 15 | 31
  White | 83 | 92 | 175
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 102 | 108 | 210
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.29 (5.619) | 29.02 (5.099) | 29.15 (5.347)
Duration of Exposure [Mean (Standard Deviation); unit: days] | 29.7 (44.28) | 33.4 (57.94) | 31.6 (51.54)
percentage of predicted FEV1 [Mean (Standard Deviation); unit: Percent] | 94.86 (18.277) | 94.99 (17.487) | 94.93 (17.832)

OUTCOME MEASURES:

1. Primary Outcome: Severity of COVID-19: Evaluation of the Severity of COVID-19 as Measured by the Maximum Difference From the Baseline Value in the OSCI Within 28 Days From the Start of Experimental Therapy.
Description: To determine the efficacy of PUL-042 Inhalation Solution in the prevention of viral infection with SARS-CoV-2 and progression to COVID-19 in subjects: 1) who have repeated exposure to individuals with SARS-CoV-2 infection and, 2) are asymptomatic at enrollment.
  The primary endpoint is the severity of COVID-19 as measured by the maximum difference from the baseline value in the Ordinal Scale for Symptom Improvement (OSCI) within 28 days from the start of experimental therapy.
  The OSCI to be used in this study is derived from a draft scale proposed by the World Health Organization for clinical improvement as presented below. The minimum score is 0, maximum is 8. Higher values represent a worse outcome.
  OSCI Scale:
  0 (no evidence of infection), 1 (infected, no limitation of activities), 2 (limitation of activities), 3 (hospitalized), 4 (hospitalized & requiring oxygen), 5 (requiring high flow oxygen), 6 (requiring mechanical ventilation), 7
Time Frame: 28 days
Population: The population analyzed is the ITT (Intent-to-Treat) population minus one participant on PUL-042 that was excluded due to an absent baseline measurement.
  ITT total: 210; ITT placebo: 108; ITT PUL-042: 102
Measure: Least Squares Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 101 | 108
score on a scale | 0.028 [-0.004 to 0.060] | 0.048 [0.017 to 0.079]

2. Secondary Outcome: Percentage of SARS-CoV-2 Infections Through Day 29
Description: Positive test for SARS-CoV-2 infection 28 days from the start of experimental therapy in subjects who test negative for SARS-CoV-2 at the pre-treatment visit.
Time Frame: 28 days
Population: Percentage of participants who had a positive result from the SARS-CoV-2 test within 28 days from the first dose of study drug was assessed using the modified ITT Set.
  Participants who had a missing test result or a result of "Indeterminate" at Day 29 and did not have a positive test result at Day 15 were excluded from the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 94 | 98
percentage of participants | 3.37 [0.92 to 8.48] | 3.23 [0.88 to 8.13]

3. Secondary Outcome: Percentage of SARS-CoV-2 Infections Through Day 15
Description: Positive test for SARS-CoV-2 infection 14 days from the start of experimental therapy in subjects who test negative for SARS-CoV-2 at the pre-treatment visit.
Time Frame: 14 days
Population: Percentage of participants who had a positive result from the SARS-CoV-2 test within 14 days from the first dose of study drug was assessed using the modified ITT Set.
  Participants who had a missing test result or a result of "Indeterminate" at Day 29 and did not have a positive test result at Day 15 were excluded from the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 94 | 98
percentage of participants | 2.17 [0.39 to 6.69] | 2.13 [0.38 to 6.55]

4. Secondary Outcome: Severity of COVID-19: Evaluation of the Severity of COVID-19 as Measured by the Maximum Difference From the Baseline Value in the OSCI Within 14 Days From the Start of Experimental Therapy.
Description: To determine the efficacy of PUL-042 Inhalation Solution in the prevention of viral infection with SARS-CoV-2 and progression to COVID-19 in subjects: 1) who have repeated exposure to individuals with SARS-CoV-2 infection and, 2) are asymptomatic at enrollment.
  The primary endpoint is the severity of COVID-19 as measured by the maximum difference from the baseline value in the Ordinal Scale for Symptom Improvement (OSCI) within 14 days from the start of experimental therapy.
  The Ordinal Scale for Clinical Improvement (OSCI) to be used in this study is derived from a draft scale proposed by the World Health Organization for clinical improvement as presented below. Higher values represent a worse outcome.
  OSCI Scale: 0 (no evidence of infection), 1 (infected, no limitation of activities), 2 (limitation of activities), 3 (hospitalized), 4 (hospitalized & requiring oxygen), 5 (requiring high flow oxygen), 6 (requiring mechanical ventilation), 7 (requiring RRT, ECMO etc.), 8 (death).
Time Frame: 14 days
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 101 | 108
score on a scale | 0.018 [-0.012 to 0.048] | 0.048 [0.019 to 0.077]

5. Secondary Outcome: Number of Participants With ICU Admission
Description: The requirement for ICU admission within 28 days from the start of experimental therapy.
Time Frame: 28 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 102 | 108
Participants | 0 | 0

6. Secondary Outcome: Number of Participants Requiring Mechanical Ventilation
Description: The requirement for mechanical ventilation within 28 days from the start of experimental therapy.
Time Frame: 28 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 102 | 108
Participants | 0 | 0

7. Secondary Outcome: Number of Participant Deaths
Description: All cause mortality at 28 days from the start of experimental therapy.
Time Frame: 28 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 102 | 108
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: full treatment period (29 days)
Description: A total of 217 participants were randomized to the study: 7 participants were randomized but not treated, 210 (96.8%) participants were included in the ITT (Intent-to-Treat) Population and Safety Population.
  Adverse events are collected by organ system, irrespective of causality.
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/108
Other Adverse Events (participants affected / at risk) | 28/102 | 10/108
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PUL-042 Inhalation Solution (N=102) | Sterile Saline for Inhalation (N=108)
Nausea (Gastrointestinal disorders) | 1 | 1
Chest discomfort (General disorders) | 2 | 0
Chills (General disorders) | 5 | 0
Fatigue (General disorders) | 1 | 1
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 2 | 0
Hypertension (Vascular disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT04313023/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT04313023/SAP_001.pdf